CLINICAL TRIAL: NCT04611685
Title: Non-Steroidal Anti-inflammatory Drugs (NSAIDS) vs. Tramadol in Pain Management After Transnasal Transsphenoidal Surgery Among Patients With Pituitary Adenomas: A Prospective Randomized Controlled Trial
Brief Title: Pain Management After Transnasal Transsphenoidal Surgery for Pituitary Adenomas
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ZS-2631
Record Dates: First submitted 2020-10-28; First posted 2020-11-02 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-11

CONDITIONS: Pituitary Adenoma; Surgery; Pain
Keywords: NSAIDs; Tramadol; Pituitary Adenoma; Pain Management; Transnasal Transsphenoidal surgery
MeSH Terms: conditions — Pituitary Neoplasms; Pain; Agnosia | interventions — Anti-Inflammatory Agents, Non-Steroidal; parecoxib; loxoprofen; Tramadol

STUDY DESIGN:
Intervention Model Description: Participants are assigned to one of two groups in parallel during the study, using the method of randomization. The ratio is 1:1.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The participant, investigator and outcome assessors are all prevented from having knowledge of the interventions assigned to individual participants. Only the care provider knows individual specified intervention.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NSAIDs (Experimental): Parecoxib (iv.) for once & Loxoprofen (po.) for routine use during the first 3 postop. days.
  Interventions: Drug: NSAID
- Tramadol (Active Comparator): Tramadol (im.) for once & Tramcontin (po.) for routine use during the first 3 postop. days.
  Interventions: Drug: Tramadol

INTERVENTIONS:
Drug: NSAID — Immediately after the operation, the patient is given (parecoxib 40 mg + sodium chloride 100 ml) intravenously once, and then given (loxoprofen 60 mg) orally twice a day during the first three postoperative days.
  Other Names: Parecoxib (iv.); Loxoprofen (po.)
  Arms: NSAIDs
Drug: Tramadol — Immediately after the operation, the patient is given (tramadol 100 mg) intramuscularly once, and then given (tramcontin 100 mg) orally twice a day during the first three postoperative days.
  Other Names: Tramadol (iv.); Tramcontin (po.)
  Arms: Tramadol

SUMMARY:
We hypothesize that the effects of non-steroidal anti-inflammatory drugs (NSAIDS) for pain relief among patients with pituitary adenomas undergoing transnasal transsphenoidal surgeries are non-inferior to tramadol. We aim to launch a single-center randomized clinical trial to verify this hypothesis.

DETAILED DESCRIPTION:
Postoperative pain is an important clinical concern and quality-of-care metric, yet it is undertreated in neurosurgical patients. Approximately 40% of inpatients complain of severe pain postoperatively, and only 56% of these patients indicate that their pain is well controlled. In addition, pain is a common cause of delayed discharge and unplanned hospital readmission.

Pituitary adenoma is the second most common benign primary central nervous system tumor, and transnasal transsphenoidal (TTS) has long taken over craniotomy to be the first-line surgical approach for pituitary tumor resection. TTS significantly reduces patient's surgical trauma, shortens the operation time, reduces surgery-related complications, and increases total tumor resection rate compared with the previously used craniotomy. However, given that the nasal mucosa is extremely sensitive, the feeling of pain is more obvious after surgery via TTS approach than via craniotomy.

Opioids such as morphine and pethidine are the most effective post-surgical analgesics, but they have a series of side effects, such as drug addiction, decreased gastrointestinal motility, nausea and vomiting. Opioids are not an analgesic that must be used after TTS surgery. NSAIDS, such as parecoxib and lexone, and tramadol are also commonly used analgesics after surgery, and they are also effective. NSAIDS is a first-tier painkiller, and tramadol is a second-tier drug. There is no evidence-based evidence recommending the preferred choice of these two drugs. Which of NSAIDS and tramadol has the better analgesic effect and which drug brings lower side effects to patients is still unclear. The clinical application of the two drugs is entirely based on the personal habits of the surgeon.

Therefore, we plan to conduct a prospective randomized controlled trial to explore: whether the analgesic effect of NSAIDS is non-inferior than tramadol; and whether the side effects of NSAIDS are not higher than tramadol. This result will guide us in clinical pain management for patients with pituitary adenomas after surgery via TTS approach.

ELIGIBILITY:
Inclusion Criteria:

* Patients with pituitary adenomas that need transnasal transsphenoidal surgery
* Patients of either gender aged 18 to 70 years

Exclusion Criteria:

* Patients with rhinitis, sinusitis, deviated nasal septum, etc. that can cause nasal pain
* Patients with medical history of digestive ulcer/gastrointestinal bleeding
* Patients with heart disease, severe liver and kidney dysfunction
* Pregnant patients
* Patients allergic to NSAIDs or tramadol
* Patients who need long-term treatment of NSAIDs or analgesic for other reasons
* Patients whose postoperative paraffin pathology suggests non-pituitary adenoma
* Patients who have not undergone transsphenoidal surgery
* Patients who reject to enter the group or ask to leave the group after entry

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Estimated)
Dates: Start 2020-10-31 (Actual); Primary Completion 2021-10 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
The VAS scores of patients | 24 hours after the surgery
  visual analogue scale score that represents the patient's subjective pain perception

SECONDARY OUTCOMES:
The VAS scores of patients | 48 hours after the surgery
  visual analogue scale score that represents the patient's subjective pain perception
The VAS scores of patients | 72 hours after the surgery
  visual analogue scale score that represents the patient's subjective pain perception
The dynamic trend of VAS scores of patients during the first 3 postoperative days | during the first 3 postoperative days
  visual analogue scale score that represents the patient's subjective pain perception

OTHER OUTCOMES:
The side effects of the drugs | during the first 3 postoperative days
  Including but not limited to nausea, vomiting, upset stomach, stomach pain, gastrorrhagia, dizziness and skin rash, while using these drugs

CONTACTS AND LOCATIONS:
Overall Officials: Bing Xing, MD, Study Chair — Neurosurgery, Peking Union Medical College Hospital, Beijing, China; Wei Lian, MD, Study Director — Neurosurgery, Peking Union Medical College Hospital, Beijing, China
Locations (1):
- Peking Union Medical College Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
The individual participant data can be made available upon reasonable request to the study chair, Dr. Bing Xing, or the study director, Dr. Wei Lian.

REFERENCES:
- [Background] Titsworth WL, Abram J, Guin P, Herman MA, West J, Davis NW, Bushwitz J, Hurley RW, Seubert CN. A prospective time-series quality improvement trial of a standardized analgesia protocol to reduce postoperative pain among neurosurgery patients. J Neurosurg. 2016 Dec;125(6):1523-1532. doi: 10.3171/2015.10.JNS15698. Epub 2016 Mar 11. PMID 26967774
- [Background] Quiney N, Cooper R, Stoneham M, Walters F. Pain after craniotomy. A time for reappraisal? Br J Neurosurg. 1996 Jun;10(3):295-9. doi: 10.1080/02688699650040179. PMID 8799542
- [Background] Joshi GP, Ogunnaike BO. Consequences of inadequate postoperative pain relief and chronic persistent postoperative pain. Anesthesiol Clin North Am. 2005 Mar;23(1):21-36. doi: 10.1016/j.atc.2004.11.013. PMID 15763409
- [Background] Shepherd DM, Jahnke H, White WL, Little AS. Randomized, double-blinded, placebo-controlled trial comparing two multimodal opioid-minimizing pain management regimens following transsphenoidal surgery. J Neurosurg. 2018 Feb;128(2):444-451. doi: 10.3171/2016.10.JNS161355. Epub 2017 Mar 3. PMID 28298041
- [Background] Molitch ME. Diagnosis and Treatment of Pituitary Adenomas: A Review. JAMA. 2017 Feb 7;317(5):516-524. doi: 10.1001/jama.2016.19699. PMID 28170483